CLINICAL TRIAL: NCT03974620
Title: Individual Placement and Support (IPS) and Cognitive Remediation Therapy (CRT) as an Adjunct to Treatment as Usual (TAU) in Patients With Early Schizophrenia Spectrum Disorder: Study Protocol for a Randomized Controlled Feasibility Trial
Brief Title: Individual Placement and Support and/or Cognitive Remediation Therapy Added to TAU in Patients With Early Schizophrenia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: PILL-IPS&CRT- 001
Record Dates: First submitted 2019-05-18; First posted 2019-06-05 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Schizophrenia; Schizophreniform Disorders; Schizoaffective Disorder; Psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Individual Placement and Support (IPS) (Experimental): IPS is a vocational support program to facilitate return to employment in individuals with severe and enduring mental illnesses.
  Interventions: Behavioral: Individual Placement and Support
- Cognitive Remediation Therapy (CRT) (Experimental): CRT will be delivered twice weekly individual computerised CRT with therapist input. This therapy will be delivered by a CRT trained assistant psychologist.
  Interventions: Behavioral: Cognitive Remediation Therapy
- IPS and CRT (Experimental): A combination of IPS and CRT will be provided to participants in this arm.
  Interventions: Behavioral: Individual Placement and Support; Behavioral: Cognitive Remediation Therapy
- Treatment as usual (No Intervention): Continued input as normal with treating psychiatrist.

INTERVENTIONS:
Behavioral: Individual Placement and Support — Individual Placement and Support is a vocational support program that was developed in the USA, to facilitate return to employment in individuals with severe and enduring mental illnesses.
  Arms: IPS and CRT; Individual Placement and Support (IPS)
Behavioral: Cognitive Remediation Therapy — This is an evidence based intervention that aims to improve cognitive functioning.
  Arms: Cognitive Remediation Therapy (CRT); IPS and CRT

SUMMARY:
This study aims to test the hypothesis that addition of Individual Placement and Support (IPS) and/or Cognitive Remediation Therapy (CRT) in addition to treatment as usual in patients with early psychosis will be feasible and acceptable in patients with early schizophrenia.

DETAILED DESCRIPTION:
This is an assessor blind, randomised controlled trial, employing a factorial design. This trial aims to assess the feasibility of IPS, CRT or their combination as an add on to treatment as usual. Patients with early schizophrenia spectrum disorder will be recruited from major psychiatric units in Pakistan. Treatment as usual (TAU) will comprise of patient's current antipsychotic medication as prescribed by their responsible clinician. Patients will be randomised into IPS, CRT, their combination or TAU, according to the 2x2 factorial schedule in the table. A total of 30 participants will be recruited in each cell, giving a total of 120 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male/Female patients aged between 18-35 years.
2. Diagnosis of schizophrenia confirmed by SCID meeting DSM-V criteria for schizophrenia, schizophreniform or schizoaffective psychosis.
3. Stable on medication for the past four weeks.
4. In contact with mental health services
5. Within 5 years of diagnosis.
6. Able to demonstrate the capacity to provide informed consent to take part in this feasibility trial, as assessed by their own clinician.

Exclusion Criteria:

1. Active DSM-V substance abuse (except nicotine or caffeine) or dependence within the last three months
2. Relevant CNS or other medical disorders
3. Diagnosis of Learning Disability.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of undertaking a trial of the intervention, as determined by: Recruitment and attrition rates | 6 month post intervention
  Recruitment and attrition rates: This will be determined using recruitment and attrition rates into the trial
Acceptability of the intervention, as determined by: number of sessions attended | 6 months post intervention
  Therapy logs: therapy logs with number of sessions attended
Client Satisfaction Questionnaire (CSQ) | 6 month post intervention
  Participants' satisfaction will be measured using CSQ-8. The scale consists of 8 items score range from 8 to 32, with higher values indicating higher satisfaction.

IPD SHARING:
Plan to Share IPD: No
Anonymised data once analysed and published will be available on reasonable request.